CLINICAL TRIAL: NCT03410420
Title: Detection of Hypoxia in Human Thoracic Aorta Using Pimonidazole Hydrochloride
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Gleason (Other)
Responsible Party: Sponsor-Investigator, Thomas Gleason, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY19090250
Record Dates: First submitted 2018-01-08; First posted 2018-01-25 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Aortic Aneurysm, Thoracic
Keywords: Thoracic Aortic Aneurysm; Hypoxia; Ascending Aorta; Hypoxyprobe; Pimonidazole
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Hypoxia

STUDY DESIGN:
Intervention Model Description: This is a prospective study designed to determine the safety and value of pimonidazole hydrochloride to detect levels of tissue hypoxia in patients presenting with ascending aortic aneurysm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Non aneurysmal (Active Comparator): Intervention: four non-aneurysmal patients undergoing coronary artery bypass graft or aortic valve replacement will be administered pimonidazole-HCl orally in a single dose (0.5g/m2) 24 hours prior to scheduled surgical time.
  Interventions: Drug: Pimonidazole hydrochloride
- Aneurysmal (Experimental): Intervention: four patients who are candidates for aortic replacement due to aneurysm will be administered pimonidazole-HCl orally in a single dose (0.5g/m2) 24 hours prior to scheduled surgical time.
  Interventions: Drug: Pimonidazole hydrochloride

INTERVENTIONS:
Drug: Pimonidazole hydrochloride — administration of pimonidazole-HCl

SUMMARY:
This is a prospective study designed to determine the safety and value of Hypoxyprobe-1 (pimonidazole hydrochloride (-HCl)) to detect levels of tissue hypoxia in patients presenting with ascending aortic aneurysm.

DETAILED DESCRIPTION:
The proposed study is designed to identify the level of tissue hypoxia in patients presenting with ascending aortic aneurysm. Ascending aortic aneurysms affect approximately 15,000 people in the United States each year, and represent a serious clinical problem because there is a known, but unspecified risk of aortic rupture or dissection. Despite progress made in the surgical management of ascending aortic aneurysms, the molecular and cellular mechanisms involved remain elusive. However, indirect evidence of tissue hypoxia have recently been described in the literature.

This pilot study will use pimonidazole-HCl, a compound that is retained by hypoxic cells and that has been used for detection of tissue hypoxia in human since the early 2000s. This pilot study will involve twenty patients who are candidates for aortic replacement due to aneurysm and twenty non-aneurysmal patients undergoing coronary artery bypass graft (controls). Patients will be administered pimonidazole-HCl orally in a single dose (0.5g/m2) 24 hours prior to scheduled surgical time. During surgery, the resected aneurysmal aortic specimens (for patients undergoing aortic replacement) or aortic punch (for patients undergoing coronary artery bypass graft) will be harvested. Tissue hypoxia will be qualitatively and quantitatively assessed in the investigator's research laboratory. Based on previous toxicological animal studies and previous use in human studies, the anticipated risk of severe or serious side effect will be relatively minimal.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age who require one of the following open surgery:

   * Ascending thoracic aorta repair due to aneurysm;
   * Aortic valve replacement due to aortic valve insufficiency;
   * Coronary artery bypass graft procedure due to coronary heart disease. Imaging CT scans and echography defining the presence of ascending aortic aneurysm will be centrally reviewed prospectively to ensure adherence to subject inclusion criteria.
2. Adequate hematologic functions:

   * White blood cells > 2500/µ;
   * Platelets > 100,000/µL;
   * Hemoglobin > 8 g/dl.
3. Adequate renal functions: serum creatinine < 2.0 mg/dl.
4. Adequate hepatic function: serum alkaline phosphatase, bilirubin, and serum glutamate oxaloacetate transaminase twice normal levels.
5. If the subject or partner is of childbearing potential, he or she must be willing to use adequate contraception (hormonal or barrier method or abstinence) from the time of screening and for a period of at least 16 weeks after procedure.
6. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form, release of medical information, and Health Insurance Portability and Accountability Act (HIPAA) documentation.
7. Female subjects of childbearing potential must have a negative serum pregnancy test at screening. human chorionic gonadotropin levels will be assessed for all women of childbearing years prior to the procedure.

Exclusion Criteria:

1. Severe septicemia or severe infection in the 4 weeks prior to study entry;
2. The subject has a baseline NIHSS > 1 or modified Rankin Scale > 1.
3. Active participation in other research therapy for cardiovascular repair/regeneration;
4. Pregnant or breastfeeding at time of screening;
5. Cardiothoracic surgery within 30 days prior to screening;
6. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Detection of pimonidazole-HCl in aortic specimens | < 1 week
  Levels of pimonidazole-HCl will be quantified in aortic specimens from patients who were administered pimonidazole-HCl prior to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Gleason, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No